CLINICAL TRIAL: NCT05373979
Title: Development and Validation of Pediatric Narcolepsy Patient Reported Outcomes Scale (PN-PROS)
Brief Title: Development and Validation of Pediatric Narcolepsy Patient Reported Outcomes Scale
Acronym: PN-PROS
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Jewish Health (Other); Geisinger Clinic (Other); The Hospital for Sick Children (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Kiran Maski, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-A00029346
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Narcolepsy; Obstructive Sleep Apnea
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Narcolepsy: Narcolepsy type 1 (NT1 or narcolepsy with cataplexy) and Narcolepsy type 2 (NT2 or narcolepsy without cataplexy)
- Obstructive Sleep Apnea: mild to moderate obstructive sleep apnea (OSA; obstructive AHI of 1-15/hour)

SUMMARY:
The purpose of this study is to test a pediatric narcolepsy patient reported outcomes tool to assess pediatric narcolepsy symptoms and their effect on daily functioning and quality of life. The goal is to develop a clinical survey that can improve the care of pediatric narcolepsy.

DETAILED DESCRIPTION:
WHO IS ELIGIBLE?

* Children and adolescents with narcolepsy between the ages of 9-17 years
* Diagnosis must be verified by a signed letter from physician in order to participate
* Participants must be able to understand the purpose of the study

PARTICIPATION DETAILS

* Upon enrollment participants will receive an email containing a link to complete HIPAA compliant online surveys about narcolepsy symptoms, quality of life, and daily function. Surveys should take no more than 30 minutes.
* One week later, some participants will receive another email with a link to complete a 10-minute follow up survey

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents ages 9-17
* Have a diagnosis of narcolepsy type 1, narcolepsy type 2, or mild to moderate obstructive sleep apnea (OSA)

Exclusion Criteria:

* A history of visual or hearing impairment
* A co-morbid neurodevelopmental disorder such as autism or schizophrenia
* No access to computer/tablet/smart phone to complete questionnaires

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients (and a parent/guardian) with an established narcolepsy type 1, narcolepsy type 2, or OSA diagnoses ages 9-17 years.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Survey Validation | 2 Years
  To evaluate the content validity and reliability of the PN-PROs item pools through a field test of the item pools in a diverse, national sample of pediatric narcolepsy patients with a comparator group of pediatric mild obstructive sleep apnea patients (9-17 years).

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Maski, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers outside of Boston Children's Hospital.